CLINICAL TRIAL: NCT05275634
Title: Effect of Different Carrier Frequencies of Interferential Current on Upper Trapezius Myofascial Trigger Points: A Randomized Controlled Trial
Brief Title: Interferential Current And Trapezius Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Samir Elsaid Mohamed, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003591
Record Dates: First submitted 2022-02-15; First posted 2022-03-11 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Upper Trapezius Trigger Points
Keywords: Interferential current; Carrier frequency; Upper trapezius; Trigger points

STUDY DESIGN:
Intervention Model Description: This trial has four groups; three experimental and one group control.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard treatment and interferential current with carrier frequency 2 KHz (Experimental): Standard treatment and interferential current with carrier frequency 2 KHz will be received three times a week for four weeks.
  Interventions: Other: Stander treatment; Device: Interferential current with carrier frequency 2 KHz
- Standard treatment and interferential current with carrier frequency 4 KHz (Experimental): Standard treatment and interferential current with carrier frequency 4 KHz will be received three times a week for four weeks.
  Interventions: Other: Stander treatment; Device: Interferential current with carrier frequency 4 KHz
- Standard treatment and interferential current with carrier frequency 8 KHz (Experimental): Standard treatment and interferential current with carrier frequency 8 KHz will be received three times a week for four weeks.
  Interventions: Other: Stander treatment; Device: Interferential current with carrier frequency 8 KHz
- Standard treatment and placebo interferential current (Placebo Comparator): Standard treatment and placebo interferential current will be received three times a week for four weeks.
  Interventions: Other: Stander treatment; Device: placebo interferential current

INTERVENTIONS:
Other: Stander treatment — Standard treatment will be (active cervical range of motion exercises, myofascial release to upper trapezius muscle and postural advices at home).
Device: Interferential current with carrier frequency 2 KHz — Interferential current treatment parameters will be as following; carrier frequency 2 KHz and beat frequency 15 Hz performed for 45 minutes per session.The intensity will be raised according to the subject's tolerance, remaining in the sensory level.
  Arms: Standard treatment and interferential current with carrier frequency 2 KHz
Device: Interferential current with carrier frequency 4 KHz — Interferential current treatment parameters will be as following; carrier frequency 4 KHz and beat frequency 15 Hz performed for 45 minutes per session.The intensity will be raised according to the subject's tolerance, remaining in the sensory level.
  Arms: Standard treatment and interferential current with carrier frequency 4 KHz
Device: Interferential current with carrier frequency 8 KHz — Interferential current treatment parameters will be as following; carrier frequency 8 KHz and beat frequency 15 Hz performed for 45 minutes per session.The intensity will be raised according to the subject's tolerance, remaining in the sensory level.
  Arms: Standard treatment and interferential current with carrier frequency 8 KHz
Device: placebo interferential current — Interferential current intensity will not be raised.
  Arms: Standard treatment and placebo interferential current

SUMMARY:
To investigate the effect of different carrier frequencies of interferential current on pressure pain threshold, neck disability, cervical range of motion and upper trapezius muscle activity when applied on upper trapezius chronic myofascial trigger points: Randomized Controlled Trial

DETAILED DESCRIPTION:
Interferential current (IFC) is a medium frequency current derived from the interference of two symmetrical, but asynchronous alternating currents ranged from 1 to 10 KHz. The two main currents resulting in a single interference current with properties uniquely different from the two original currents.The lesser current of the two original currents is termed the carrier frequency and the interference current is called the beat frequency. A specific beat frequency can be obtained from several possible interference currents as long as the difference between the original currents is the same. For electro pain modulation, IFC is commonly used form of electrotherapy. It has the advantage of reducing the skin impedance, deeper penetration into tissues and is perceived as more comfortable.

Myofascial pain syndrome (MPS) is a common form of chronic musculoskeletal pain that widely spread and contributing to a significant financial burden and job- related disability. It represents the most common disorder in patients with nonspecific chronic neck pain.The main characteristics of MPS include the presence of myofascial trigger points (MTrPs) which are defined as hyperirritable nodule in a taut band of skeletal muscle fibers which is palpable and tender during physical examination. Trigger points (TrPs) are usually seen in the upper fiber of trapezius. TrPs can be clinically classified as either active or latent. Active TrPs was defined as: MTrPs that refer pain during activity and during rest without any pressure. They prevent full muscle lengthening and induce their weakness. Latent TrPs was defined as: MTrPs that is painful only when palpated. Evidence on the effect of IFC on pain modulation is not confirmed up till now. This might be attributed to multiple factors such as limited number of studies, inappropriate use of the parameters or using single carrier frequency (4 KHz) in majority of studies and the physiological effects of all our modalities are dose dependent. Dose depends on details of parameters including frequency. For IFC, the carrier frequency of the current has been suggested as an important parameter to achieve the most effective hypoalgesic response. However, there remains no evidence to support the selection of one carrier frequency over another. Few studies were conducted to examine the effect of different carrier frequencies by comparing their individual effects. Further researches are needed to prove which carrier frequency is more effective in treatment. Therefore, this study will be conducted to compare the effect of different carrier frequencies of the IFC in the management of upper trapezius chronic TrPs.

ELIGIBILITY:
Inclusion Criteria:

* Ages from18-29 years old with unilateral chronic myofascial trigger points in upper trapezius muscle will be included in this study.
* Participants have chronic myofascial trigger points if they have pain with pressure, local twitch response, jump sign, limited range of motion and referred pain lies over the lateral aspect of the upper trapezius fibers and superiorly to the ipsilateral occiput.
* Normal body mass index (BMI) from 18-24.9 Kg/m (BMI = body mass in kg divided by participant height in meters).

Exclusion Criteria:

* Onset of pain less than 3 months
* History of whiplash injury
* History of cervical spine surgery
* Cervical radiculopathy or myelopathy and cervical disc lesion
* Cervical spondylolisthesis
* Having multiple sclerosis, thyroid dysfunction and chronic infection
* Having rheumatologic condition as poly articular osteoarthritis, rheumatoid arthritis and advanced cervical spine degenerative diseases
* Skin disease and impaired sensation
* Phobia of using electrical current
* Pregnancy, tumor, thrombosis and pacemaker
* Administration of regular analgesic drugs or any medications that affect skin sensation.
* Receiving physical therapy intervention during the past three months.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain threshold | Immediately after the end of the treatment
  Pressure pain threshold will be measured by digital pressure algometer

SECONDARY OUTCOMES:
Change in Pressure pain threshold | 12 weeks following the end of the treatment
  Pressure pain threshold will be measured by digital pressure algometer
Change in neck disability | Immediately after the end of the treatment
  Neck disability will be measured by Arabic neck disability index
Change in neck disability | 12 weeks following the end of the treatment
  Neck disability will be measured by Arabic neck disability index
Change in cervical range of motion | Immediately after the end of the treatment
  Cervical range of motion will be measured by cervical range of motion device
Change in cervical range of motion | 12 weeks following the end of the treatment
  Cervical range of motion will be measured by cervical range of motion device
Change in upper trapezius muscle activity | Immediately after the end of the treatment
  Muscle activity will be measured by electromyography in the form of root mean square
Change in upper trapezius muscle activity | 12 weeks following the end of the treatment
  Muscle activity will be measured by electromyography in the form of root mean square

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt

REFERENCES:
- [Background] Venancio RC, Pelegrini S, Gomes DQ, Nakano EY, Liebano RE. Effects of carrier frequency of interferential current on pressure pain threshold and sensory comfort in humans. Arch Phys Med Rehabil. 2013 Jan;94(1):95-102. doi: 10.1016/j.apmr.2012.08.204. Epub 2012 Aug 23. PMID 22922327
- [Background] Correa JB, Costa LO, Oliveira NT, Lima WP, Sluka KA, Liebano RE. Effects of the carrier frequency of interferential current on pain modulation and central hypersensitivity in people with chronic nonspecific low back pain: A randomized placebo-controlled trial. Eur J Pain. 2016 Nov;20(10):1653-1666. doi: 10.1002/ejp.889. Epub 2016 May 6. PMID 27150263